CLINICAL TRIAL: NCT04019977
Title: Effects of Early Community Services on Child and Family Development
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The COVID-19 pandemic halted research activities at the collaborating hospital.
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: LifeBridge Health (Other)
Responsible Party: Principal Investigator, Lisa Berlin, Associate Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HP-00076256
Record Dates: First submitted 2019-07-12; First posted 2019-07-15 (Actual); Results first posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-01

CONDITIONS: Child Development
Keywords: Nurse Home Visiting

STUDY DESIGN:
Who Masked: Participant
Masking Description: As described above, the nurse home visiting program is being provided on a random-assignment basis according to child birthdate. Nurse home visitors will enroll new mothers into the nurse home visiting program every other day only (on odd dates). The new mothers who give birth on an even date will not be offered the nurse home visiting program. They will be considered the "control" group and are expected to access community services as they normally would.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nurse Home Visiting Group (Experimental): This group will be offered services from the nurse home visiting program.
  Interventions: Other: Nurse Home Visiting Program
- Non-intervention Group (No Intervention): This group will not be offered services from the nurse home visiting program.

INTERVENTIONS:
Other: Nurse Home Visiting Program — Brief nurse home visiting program
  Arms: Nurse Home Visiting Group

SUMMARY:
The purpose of the current study is to evaluate the effects on early child development of early community services, including a brief nurse home visiting program. Investigators hypothesize that nurse home visiting program participants will be significantly different than non- nurse home visiting program participants on the following child and family outcomes: (a) (reduced) infant emergency room use and overnight hospital stays; (b) (increased) family use of community resources and (higher quality) child care; (c) (increased) maternal wellbeing; and (d) (increased) quality of the home environment, including home safety and supportive parenting by both parents. The study will also explore long-term differences between the nurse home visiting program recipients and non-recipients in (a) rates of official investigations for child maltreatment and (b) two indicators of early educational achievement: kindergarten readiness scores and rates of kindergarten attendance.

DETAILED DESCRIPTION:
The purpose of the current study is to evaluate the effects on child and family development of early community services, including a brief nurse home visiting program. The proposed study will be conducted in partnership with the brief nurse home visiting program and Sinai Hospital, both located in Baltimore, MD. For the purposes of this study, Sinai Hospital will serve as the community/catchment area. Nurse home visitors enroll new mothers into the nurse home visiting program while they are still in the hospital/maternity ward. When the current study officially begins, nurse home visitors will recruit new mothers into the nurse home visiting program every other day only (on odd dates). Research staff will recruit all Baltimore City residents who give birth at Sinai Hospital, regardless of odd/even birth date, while they are still in the hospital/maternity ward.

ELIGIBILITY:
Inclusion Criteria:

* Mother and Infant are Baltimore City Residents
* Mother gave birth to infant at Sinai Hospital in Baltimore, MD beginning approximately July 15, 2019
* Mother speaks English

Exclusion Criteria:

* Mother and Infant are not Baltimore City Residents
* Mother did not give birth to infant at Sinai Hospital in Baltimore, MD beginning approximately July 15, 2019
* Mother does not speak English

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 277 (Actual)
Dates: Start 2019-07-18 (Actual); Primary Completion 2020-09-29 (Actual); Study Completion 2021-07-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa J Berlin, PhD, Principal Investigator — University of Maryland
Locations (2):
- United States (2):
  - UMaryland, Baltimore, Maryland
  - Sinai Hospital, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No
Individual results will not be shared with participants nor their primary care physician. Study results will be shared in aggregate in the form of a one-page infographic available to study participants at their request. De-identified and masked study findings will be shared with the Sinai Hospital research team and with other community service providers upon request. Finally, aggregate findings will be reported in scholarly journals.

REFERENCES:
- [Background] Dodge KA, Goodman WB, Murphy RA, O'Donnell K, Sato J. Randomized controlled trial of universal postnatal nurse home visiting: impact on emergency care. Pediatrics. 2013 Nov;132 Suppl 2(Suppl 2):S140-6. doi: 10.1542/peds.2013-1021M. PMID 24187116
- [Background] Dodge KA, Goodman WB, Murphy RA, O'Donnell K, Sato J, Guptill S. Implementation and randomized controlled trial evaluation of universal postnatal nurse home visiting. Am J Public Health. 2014 Feb;104 Suppl 1(Suppl 1):S136-43. doi: 10.2105/AJPH.2013.301361. Epub 2013 Dec 19. PMID 24354833

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From July 2019-March 2020, FCM staff recruited the treatment group: City residents who gave birth at a local hospital on odd dates. Simultaneously, research staff invited all city residents who gave birth at this Hospital as the control group. However, due to COVID-19, participants in the treatment group did not receive nurse visits as planned and recruitment abruptly stopped in March 2020.
Pre-assignment Details: Due to the COVID-19 pandemic and the participating hospital halting research activities, recruitment abruptly stopped in March, 2020, and participants in the treatment group did not receive the intervention. Because randomization and service delivery failed to occur, results are reported as an aggregate of all 152 participants that completed an interview.
Groups:
- Completed Interview: Participants who gave birth at Hospital, were City residents, enrolled in the study and completed the interview.
Period: Overall Study
Arm/Group | Completed Interview
Started | 152
Completed | 152
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Enrolled participants who completed the cross-sectional interview
Groups:
- Completed Interview: The mothers enrolled in the study and completed the interview.
Arm/Group | Completed Interview
Number analyzed (Participants) | 152
Age, Continuous [Mean (Full Range); unit: years] | 29.87 [18 to 42]
Sex: Female, Male [Count of Participants; unit: Participants] — Interview
  Participants
    Female | 152
    Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Interview
  Participants
    Hispanic or Latino | 5
    Not Hispanic or Latino | 146
    Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 71
  White | 71
  More than one race | 6
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Study-specific Structured Maternal Report Interview on Infant Emergency Room Use
Description: maternal report of infant emergency room use during study-specific structured interview, i.e.: Since you came home from the hospital after birth, has the baby had to go to the emergency room or emergency department for an illness, injury, or emergency?
Time Frame: collected at/around the time infant turned 6 months old (approximately 6 months from baseline); Due to COVID-related disruptions, we loosened time parameters to anytime we could reach the family; Mean age = 6.78 m; Acceptable/actual range= 5.8-14 m
Population: Those who completed the interview
Measure: Count of Participants; unit: Participants
Groups:
- Infant ER Visit: If the infant has visited the ER, and if so, how many times.
Arm/Group | Infant ER Visit
Number analyzed (Participants) | 152
Participants
  Yes | 20
  No | 132

2. Primary Outcome: Data Collection From Records on Infant Emergency Room Use
Description: records from Sinai Hospital and/or the Maryland Department of Health indicating number of emergency room visits
Time Frame: Intended collection time: five and a half years post-psychosocial interview; Unable to collect due to study termination
Population: Due to COVID-19, this study ended prematurely, in March 2020. No follow-up interview was conducted.
Arm/Group | Infant ER Visit
Number analyzed (Participants) | 0

3. Primary Outcome: Study-specific Structured Maternal Report Interview on Number of Infant Overnight Hospital Stays
Description: maternal report of number of infant overnight hospital stays during study-specific structured interview, i.e.: Since you came home from the hospital after birth, has the baby stayed overnight in the hospital for an illness, injury, or emergency? If yes, how many times?
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Infant ER Visit
Number analyzed (Participants) | 152
Participants
  Yes | 7
  No | 145

4. Primary Outcome: Data Collection From Records on Infant Overnight Hospital Stays
Description: records from Sinai Hospital and/or the Maryland Department of Health indicating number of overnight hospital stays
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: number of overnight hospital stays
Arm/Group | Completed Interview
Number analyzed (Participants) | 152
number of overnight hospital stays | 0.05 (0.21)

5. Primary Outcome: Study-specific Structured Maternal Report Interview on Family Use of Community Resources
Description: Mothers were asked if they use the following services (yes/no): Food Stamps, Special Supplemental Nutrition Program for Women, Infants and Children (WIC), Supplemental Security Income (SSI), Work First- Family Cash Assistance, Medicaid (for the mother) or State Children's Health Insurance Program (S-CHIP) for child, Private health insurance, Job seeking assistance, Transportation assistance, Shelter/housing assistance, Food assistance, Clothing assistance, Furniture assistance, Heating/cooling assistance, Family planning clinic, Breastfeeding support, Mental health counseling, Substance use support, Couples counseling or domestic violence help, Veterans Affairs, Child Protective Services (CPS), Faith-based services, Maryland Family Network, The ARC of Maryland (for disabilities), B'more for Healthy Babies (services to prevent infant mortality), child care subsidy service, child care center or home based child care with other children or individual child care provider, Other
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Number of resources used
Arm/Group | Completed Interview
Number analyzed (Participants) | 152
Number of resources used | 3.99 (2.24)

6. Primary Outcome: Study-specific Structured Maternal Report Interview on Family Use of Community Resources (Cont.)
Description: as for outcome 5
Time Frame: as for outcome 1
Population: Total n's may be less than 152 due to missing data.
Measure: Count of Participants; unit: Participants
Arm/Group | Completed Interview
Number analyzed (Participants) | 152
Participants
  SNAP: yes | 61
  SNAP: no | 91
  WIC: yes | 89
  WIC: no | 63
  SSI: yes | 2
  SSI: no | 150
  TCA: yes | 17
  TCA: no | 135
  Medicaid: yes | 75
  Medicaid: no | 77
  SCHIP: yes | 96
  SCHIP: no | 56
  Private health insurance: yes | 74
  Private health insurance: no | 78
  Job services: yes | 7
  Job services: no | 145
  Transportation assistance: yes | 4
  Transportation assistance: no | 148
  Shelter assistance: yes | 0
  Shelter assistance: no | 152
  Housing assistance: yes | 3
  Housing assistance: no | 149
  Food bank: number analyzed (Participants) | 151
  Food bank: yes | 9
  Food bank: no | 142
  Clothing assistance: yes | 3
  Clothing assistance: no | 149
  Furniture assistance: yes | 0
  Furniture assistance: no | 152
  Heating/cooling assistance: yes | 2
  Heating/cooling assistance: no | 150
  Family planning clinic: number analyzed (Participants) | 150
  Family planning clinic: yes | 3
  Family planning clinic: no | 147

7. Primary Outcome: Maternal Wellbeing as Assessed Using the Parenting Stress Index
Description: During the study-specific structured interview, maternal stress was measured using the Parenting Stress Index-Short Form (PSI-SF), which includes three subscales-Parental Distress, Parent-Child Dysfunctional Interaction, and Difficult Child, each containing 12 items. Mothers rated each of the 36 items on a 5-point scale ranging from strongly disagree (1) to strongly agree (5). Subscales are summed to compute a total score. The possible range is 36-180. Higher raw scores generally indicate higher levels of stress.
Time Frame: as for outcome 1
Population: 3 participants did not respond to this question
Measure: Mean (Standard Deviation); unit: total score on a scale
Arm/Group | Completed Interview
Number analyzed (Participants) | 149
total score on a scale | 53.56 (19.59)

8. Primary Outcome: Maternal Social Support as Assessed Using The Social Provisions Scale
Description: Maternal social support was assessed using The Social Provisions Scale during study-specific structured interview. Mothers were asked to think about their current relationships and rate 24 statements on a scale of 1 (strongly disagree) to 4 (strongly agree). The possible total range is 12-48, with higher scores indicating higher levels of social support.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: total score on a scale
Arm/Group | Completed Interview
Number analyzed (Participants) | 152
total score on a scale | 44.26 (5.07)

9. Primary Outcome: Maternal Wellbeing as Assessed Using the Edinburgh Postpartum Depression Scale
Description: maternal wellbeing as assessed using Edinburgh Postpartum Depression Scale (EPDS) during study-specific structured interview
  The possible range for the EPDS is 0-30, with higher scores indicating more depressive symptoms. Scores greater than or equal to 13 indicate possible clinical depression.
Time Frame: as for outcome 1
Population: N does not equal 152 due to missing data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Completed Interview
Number analyzed (Participants) | 151
units on a scale | 4.72 (3.93)

10. Primary Outcome: Maternal Wellbeing as Assessed Using the Generalized Anxiety Disorder (GAD-7)
Description: During the study-specific structured interview, maternal well-being was measured using the Generalized Anxiety Disorder (GAD-7). Mothers were asked seven questions about how often they have been bothered by various problems, on a scale from 0 (not at all) to 3 (nearly every day). If they checked off any problems, they were additionally asked how difficult the problems have made it for them to do work, take care of things, or get along with others, on a scale from 0 (not difficult at all) to 3 (nearly every day).The possible range is a total score of 0-24, with higher scores indicating greater anxiety.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: total score on a scale
Arm/Group | Completed Interview
Number analyzed (Participants) | 152
total score on a scale | 4.01 (3.53)

11. Primary Outcome: Maternal Wellbeing as Assessed Using Study-specific Structured Interview on Health Status
Description: maternal wellbeing as assessed using study-specific structured interview, i.e.: Are you or your partner using any form of contraception or birth control at this time? Since you came home from the hospital after birth, have you had to go to your doctor or a health clinic, to the emergency room or emergency department, or stayed overnight in the hospital for illness/injury/emergency? Did you complete your 6-week post-partum check-up? Do you currently have any kind of chronic health conditions? If yes, are you under the regular care of a doctor to help manage this condition? What type of health care provider do you regularly see? In general, how do you pay for your health care? If you were sick and you wanted to be seen by a doctor, where would you go for care?
Time Frame: as for outcome 1
Population: Participants did not respond to all questions and each row represents another outcome related to the main outcome.
Measure: Count of Participants; unit: Participants
Groups:
- Maternal Wellbeing: Not all participants responded to this question.
Arm/Group | Maternal Wellbeing
Number analyzed (Participants) | 152
Participants
  Dr. or clinic visit(s) for mother illness, injury, or emergency: Yes | 51
  Dr. or clinic visit(s) for mother illness, injury, or emergency: No | 101
  Dr. or clinic visit(s) for mother illness, injury, or emergency: Refused or N/A | 0
  Completed maternal 6-week post-partum check-up: Yes | 142
  Completed maternal 6-week post-partum check-up: No | 10
  Completed maternal 6-week post-partum check-up: Refused or N/A | 0
  Chronic health conditions such as high blood pressure or diabetes: number analyzed (Participants) | 151
  Chronic health conditions such as high blood pressure or diabetes: Yes | 21
  Chronic health conditions such as high blood pressure or diabetes: No | 130
  Chronic health conditions such as high blood pressure or diabetes: Refused or N/A | 0
  Sees a health care provider regularly: Yes | 125
  Sees a health care provider regularly: No | 27
  Sees a health care provider regularly: Refused or N/A | 0
  Use of contraception or birth control at this time: number analyzed (Participants) | 150
  Use of contraception or birth control at this time: Yes | 100
  Use of contraception or birth control at this time: No | 44
  Use of contraception or birth control at this time: Refused or N/A | 6
  Mother ER visits: Yes | 24
  Mother ER visits: No | 128
  Mother ER visits: Refused or N/A | 0
  Hospital overnight for mother illness, injury, or emergency: Yes | 8
  Hospital overnight for mother illness, injury, or emergency: No | 144
  Hospital overnight for mother illness, injury, or emergency: Refused or N/A | 0
  If sick and wanted to be seen by a doctor, mother would go to...PCP: Yes | 109
  If sick and wanted to be seen by a doctor, mother would go to...PCP: No | 43
  If sick and wanted to be seen by a doctor, mother would go to...PCP: Refused or N/A | 0
  If sick and wanted to be seen by a doctor, mother would go to...health care clinic/urgent care: Yes | 27
  If sick and wanted to be seen by a doctor, mother would go to...health care clinic/urgent care: No | 125
  If sick and wanted to be seen by a doctor, mother would go to...health care clinic/urgent care: Refused or N/A | 0
  If sick and wanted to be seen by a doctor, mother would go to...emergency room: Yes | 10
  If sick and wanted to be seen by a doctor, mother would go to...emergency room: No | 142
  If sick and wanted to be seen by a doctor, mother would go to...emergency room: Refused or N/A | 0
  If sick and wanted to be seen by a doctor, mother would go to...(Other): Yes | 6
  If sick and wanted to be seen by a doctor, mother would go to...(Other): No | 146
  If sick and wanted to be seen by a doctor, mother would go to...(Other): Refused or N/A | 0
  Payment for health care: out of pocket: Yes | 2
  Payment for health care: out of pocket: No | 150
  Payment for health care: out of pocket: Refused or N/A | 0
  Payment for health care: health insurance: Yes | 78
  Payment for health care: health insurance: No | 74
  Payment for health care: health insurance: Refused or N/A | 0
  Payment for health care: Medicaid: Yes | 68
  Payment for health care: Medicaid: No | 84
  Payment for health care: Medicaid: Refused or N/A | 0
  Payment for health care: Other: Yes | 4
  Payment for health care: Other: No | 148
  Payment for health care: Other: Refused or N/A | 0

12. Primary Outcome: Home Safety as Assessed Using H.O.M.E.
Description: The Home Observation for Measurement of Environment (HOME) Inventory is an observational instrument of 45 items that measures a child's home environment, including the emotional and verbal responsivity of the mother, acceptance of the child, organization of the environment, provision of appropriate play materials, maternal involvement with the child, and variety in daily stimulation.
Time Frame: Planned collection: at/around the time infant turned 6 months old; As this is an in-home observational measure only and all in-home data collection was halted due to COVID-related precautions, we do not have data for the H.O.M.E.
Population: Due to COVID-19 precautions, we did not collect these data.
Arm/Group | Completed Interview
Number analyzed (Participants) | 0

13. Primary Outcome: Home Quality as Assessed Using H.O.M.E.
Description: home quality as assessed using H.O.M.E. during study-specific structured interview
Time Frame: Planned collection: at/around the time infant turned 6 months old; As this is an in-home measure only and all in-home data collection was halted due to COVID-related precautions, we do not have data for the H.O.M.E.
Population: Due to COVID-19 precautions, we did not collect these data.
Arm/Group | Completed Interview
Number analyzed (Participants) | 0

14. Primary Outcome: Study-specific Structured Maternal Report Interview on Father's Supportive Parenting
Description: maternal report of father's supportive parenting during study-specific structured interview, i.e.: How frequently does the father/partner (with/to the baby): Play games? Sing songs or nursery rhymes? Read stories? Tell stories? Play inside with toys? Take the baby to visit relatives? Helps the baby get dressed? Feeds the baby? Hug or show physical affection to the baby? Put the baby to bed? How often does he look after the baby? How often does he run errands for you? How often does he fix things around your home, paint, or help make it look nicer in other ways? How often does he take the baby places the baby needs to go? How often does your child's father buy the following items: clothes, toys, medicine, child care items, food or formula, anything else?
Time Frame: as for outcome 1
Population: 42 mothers did not respond
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Completed Interview
Number analyzed (Participants) | 110
units on a scale | 20.94 (9.21)

15. Primary Outcome: Parenting Indicators (Discipline)
Description: 4 items to measure parental use of discipline (yes/no), type of physical punishment used (spank/tap)
Time Frame: as for outcome 1
Population: N's may not add up to 152 due to missing data
Measure: Count of Participants; unit: Participants
Arm/Group | Completed Interview
Number analyzed (Participants) | 152
Participants
  Use of physical discipline: number analyzed (Participants) | 150
  Use of physical discipline: Yes | 2
  Use of physical discipline: No | 148
  If yes, type of physical punishment used: spank/pop or slap: number analyzed (Participants) | 2
  If yes, type of physical punishment used: spank/pop or slap: Yes | 1
  If yes, type of physical punishment used: spank/pop or slap: No | 1
  If yes, type of physical punishment used: Tap: number analyzed (Participants) | 2
  If yes, type of physical punishment used: Tap: Yes | 1
  If yes, type of physical punishment used: Tap: No | 1

16. Primary Outcome: Study-specific Structured Maternal Report Interview on Quality Rating of Child's Care Center of Child Care, According to the EXCELS Rating System
Description: maternal report of quality of child care during study-specific structured interview, according to the EXCELS rating system. EXCELS is the state's child care quality rating system for all licensed family and center-based child care providers in Maryland. Programs are rated on a 1 to 5 scale according to multiple quality indicators, including developmentally appropriate learning and practice, accreditation and rating scales, licensing and compliance, staff qualifications and professional development, administrative policies, etc. Higher numbers reflect higher overall quality of the child care program.
Time Frame: as for outcome 1
Population: Only those who indicated their child is in family day care or a child care center were asked to complete this question. N's do not add to 17 due to missing data.
Measure: Count of Participants; unit: Participants
Arm/Group | Completed Interview
Number analyzed (Participants) | 15
Participants
  EXCELS Level 1 | 0
  EXCELS Level 2 | 0
  EXCELS Level 3 | 0
  EXCELS Level 4 | 2
  EXCELS Level 5 | 1
  Level unknown | 12

17. Primary Outcome: Study-specific Structured Maternal Report Interview on Infant Immunizations
Description: maternal report of infant being up to date on immunizations during study-specific structured interview, i.e. "Is the baby up to date on his/her immunizations?" (yes/no)
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Completed Interview
Number analyzed (Participants) | 152
Participants
  Yes | 138
  No | 14

18. Primary Outcome: Study-specific Structured Maternal Report Interview on Infant Well-baby Visits
Description: maternal report of infant having their well-baby visit during study-specific structured interview, i.e. "When was the last time you took the baby to see the doctor for a general examination (also known as a "well-baby visit')?" They were asked to select from the following options: within the last month, within the last three months, more than three months ago, I don't remember, I don't take my baby to the doctor for general examinations
Time Frame: as for outcome 1
Population: N's may not add to 152 due to missing data.
Measure: Count of Participants; unit: Participants
Arm/Group | Completed Interview
Number analyzed (Participants) | 152
Participants
  Within the last month | 72
  Within the last 3 months | 75
  More than 3 months ago | 5

19. Primary Outcome: Study-specific Structured Maternal Report Interview on the Number of Community Resources Family Uses
Description: maternal report of number of resources used during study-specific structured interview, i.e. a sum of all of the resources named in the interview
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: total number of resources used
Arm/Group | Completed Interview
Number analyzed (Participants) | 152
total number of resources used | 3.99 (2.24)

20. Primary Outcome: Infant Wellbeing Assessed Using Study-specific Structured Interview on Infant Health Status
Description: infant wellbeing as assessed using study-specific structured interview, i.e.: Are you currently breastfeeding? In no about how old was baby when you stopped breastfeeding? Does baby have a regular bedtime? Does baby have a regular bedtime routine? In which one position do you most often lay your baby down to sleep now? How often does baby sleep in the same bed with you or anyone else? Does anyone who lives in your home smoke cigarettes, cigars, pipes, or e-cigarettes anywhere in inside your home? Does your baby have a healthcare provider whom s/he sees regularly? If baby was sick and you wanted him/her to be seen by a doctor, where would you take baby for care? In general, how do you pay for your baby's health care?
Time Frame: as for outcome 1
Population: Multiple outcomes are measured for infant wellbeing. Therefore, not all outcomes add up to N = 152
Measure: Count of Participants; unit: Participants
Arm/Group | Completed Interview
Number analyzed (Participants) | 152
Participants
  Currently breastfeeding: yes | 138
  Currently breastfeeding: no | 14
  Infant has a regular bedtime: number analyzed (Participants) | 151
  Infant has a regular bedtime: yes | 124
  Infant has a regular bedtime: no | 27
  Infant has regular bedtime routine: number analyzed (Participants) | 151
  Infant has regular bedtime routine: yes | 138
  Infant has regular bedtime routine: no | 13
  Smoking in household: yes | 2
  Smoking in household: no | 150
  Does the baby have a healthcare provider: number analyzed (Participants) | 150
  Does the baby have a healthcare provider: yes | 148
  Does the baby have a healthcare provider: no | 2

21. Secondary Outcome: Data Collection From Records of Rates of Official Investigations for Child Maltreatment
Description: records from the Maryland Department of Human Services
Time Frame: Intended collection time: five and a half years post-psychosocial interview; Unable to collect due to study termination
Population: Due to COVID-19, this study ended prematurely, in March 2020. No follow-up interview nor record scanning was conducted.
Arm/Group | Completed Interview
Number analyzed (Participants) | 0

22. Secondary Outcome: Maternal Wellbeing as Assessed Using the Adult Attachment Style (AAS)
Description: In the AAS, mothers selected one of three brief narrative descriptions, each of which corresponds to an adult attachment style. i.e. : 1) somewhat uncomfortable being close to and trusting others …(avoidant); 2) relatively easy to get close to others and comfortable depending on them.... (secure); 3) others are reluctant to get as close as I would like (anxious)....
Time Frame: as for outcome 1
Population: 151 participants responded to this scale
Measure: Count of Participants; unit: Participants
Arm/Group | Completed Interview
Number analyzed (Participants) | 151
Participants
  Avoidant | 26
  Secure | 118
  Anxious | 7

23. Secondary Outcome: Maternal Wellbeing as Assessed Using the Adverse Childhood Experiences (ACEs)
Description: maternal wellbeing as assessed using the Adverse Childhood Experiences (ACEs) during study-specific structured interview. The range is 0-10 ACEs total.
Time Frame: as for outcome 1
Population: Total number of ACE's (0 - 10)
Measure: Mean (Standard Deviation); unit: Total ACEs
Arm/Group | Completed Interview
Number analyzed (Participants) | 144
Total ACEs | 1.5 (2.12)

24. Secondary Outcome: Neighborhood Quality as Assessed Using The Neighborhood Collective Efficacy
Description: neighborhood quality as assessed using The Neighborhood Collective Efficacy during study-specific structured interview
Time Frame: as for outcome 1
Population: (possible range 4-16)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Completed Interview
Number analyzed (Participants) | 141
units on a scale | 6.85 (2.96)

25. Secondary Outcome: Study-specific Structured Maternal Report Interview on Transportation
Description: study-specific structured maternal report interview on transportation. Participants were asked the following questions: Does anyone in your household own a working car, van, or truck? How do you usually get around, for example if you need to go somewhere like to work, the store or the doctor's office? How easy is it for you to get where you need to go (work, store, doctor's office, etc.) by personal car?
Time Frame: as for outcome 1
Population: N's may not add to 152 due to missing data.
Measure: Count of Participants; unit: Participants
Arm/Group | Completed Interview
Number analyzed (Participants) | 152
Participants
  Does anyone in the household own a working car, van, truck?: number analyzed (Participants) | 150
  Does anyone in the household own a working car, van, truck?: Yes | 138
  Does anyone in the household own a working car, van, truck?: No | 12
  Forms of transportation used: own (family) car: Yes | 122
  Forms of transportation used: own (family) car: No | 30
  Forms of transportation used: other (family) person's car: Yes | 2
  Forms of transportation used: other (family) person's car: No | 150
  Forms of transportation used: own (family) car/taxi or rideshare: Yes | 4
  Forms of transportation used: own (family) car/taxi or rideshare: No | 148
  Forms of transportation used: own (family) car/public transportation: Yes | 2
  Forms of transportation used: own (family) car/public transportation: No | 150
  Forms of transportation used: own (family) car/walk: Yes | 2
  Forms of transportation used: own (family) car/walk: No | 150
  Forms of transportation used: Other person's car: Yes | 7
  Forms of transportation used: Other person's car: No | 145
  Forms of transportation used: walk/taxi or rideshare: Yes | 5
  Forms of transportation used: walk/taxi or rideshare: No | 147
  Forms of transportation used: other person's car/public transportation: Yes | 1
  Forms of transportation used: other person's car/public transportation: No | 151
  Forms of transportation used: other person's car/public transit/CASA worker: Yes | 1
  Forms of transportation used: other person's car/public transit/CASA worker: No | 151
  Forms of transportation used: taxi/rideshare: Yes | 3
  Forms of transportation used: taxi/rideshare: No | 149
  Forms of transportation used: Public transportation: Yes | 3
  Forms of transportation used: Public transportation: No | 149
  How easy is it to get where you need to go? -- Very easy: Yes | 125
  How easy is it to get where you need to go? -- Very easy: No | 27
  How easy is it to get where you need to go?- Somewhat easy: Yes | 20
  How easy is it to get where you need to go?- Somewhat easy: No | 132
  How easy is it to get where you need to go?-- Moderately easy/difficult: Yes | 5
  How easy is it to get where you need to go?-- Moderately easy/difficult: No | 147
  How easy is it to get where you need to go?-- extremely difficult: Yes | 2
  How easy is it to get where you need to go?-- extremely difficult: No | 150

26. Other Pre Specified Outcome: Data Collection From Records of Early Educational Achievement: Kindergarten Readiness Scores, Exploratory
Description: records from the Maryland State Department of Education, exploratory
Time Frame: Intended collection time: five and a half years post-psychosocial interview; Unable to collect due to study termination
Population: We did not collect these data.
Arm/Group | Completed Interview
Number analyzed (Participants) | 0

27. Other Pre Specified Outcome: Data Collection From Records of Early Educational Achievement: Rates of Kindergarten Attendance, Exploratory
Description: records from the Maryland State Department of Education, exploratory
Time Frame: Intended collection time: five and a half years post-psychosocial interview; Unable to collect due to study termination
Population: We did not collect these data.
Arm/Group | Completed Interview
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were not assessed in this study
Description: Adverse events were not assessed in this study
Groups:
- No Adverse Events Were Monitored: No adverse events were monitored
Arm/Group | No Adverse Events Were Monitored
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-03-24): https://cdn.clinicaltrials.gov/large-docs/77/NCT04019977/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-24): https://cdn.clinicaltrials.gov/large-docs/77/NCT04019977/SAP_001.pdf